CLINICAL TRIAL: NCT03753698
Title: A Prospective, Single Arm, Interventional, Self-controlled Pilot Study to Assess the Performance and Safety of the New Generation, Wireless, Implantable Tibial Nerve Stimulator System (eCoin™) for the Treatment of Refractory Lower Urinary Tract Symptoms in Patients With Multiple Sclerosis
Brief Title: Wireless, Implantable Tibial Nerve Stimulator System (eCoin™) for the Treatment of Refractory Lower Urinary Tract Symptoms in Patients With MS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Substantial amendment to be implemented using another device
Sponsor: Chiara Zecca (Other)
Responsible Party: Sponsor-Investigator, Chiara Zecca, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EOC.NEUUR.1801
Record Dates: First submitted 2018-11-15; First posted 2018-11-27 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Lower Urinary Tract Symptoms; Posterior tibial nerve stimulation; Neuromodulation
MeSH Terms: conditions — Multiple Sclerosis; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eCoin (Experimental): Neuromodulation of posterior tibial nerve
  Interventions: Device: eCoin

INTERVENTIONS:
Device: eCoin — Implantation of device electrodes subcutaneous in lower tibia area;
  Stimulation of posterior tibial nerves:
  Regimen 1 (months 0-3): Six stimulation treatments per week, one stimulation per day, for duration of 30 minutes each Regimen 2 (months 3-6): Three stimulation treatments per week, one stimulation per day, for duration of 30 minutes each. Stimulation is activated by the patient.

SUMMARY:
Prevalence of lower urinary tract symptoms (LUTS) in patients with MS increases with disease duration. Current management of urinary clinical symptoms in MS is mainly conservative. Its long-term outcome is often poor because of the progressive disease course and the treatment related side effects. Alternative therapeutic options are botulinum toxin injections, electrical stimulation of dorsal penile/clitoral nerve, and sacral nerve modulation. Posterior tibial nerve stimulation (PTNS) is a second minimally-invasive method of electrical stimulation. Multiple benefits may derive from the development and validation of a dedicated protocol of a new self-activated neuromodulation therapy, which may improve therapy compliance/effectiveness, quality of life and social life in MS patients with refractory LUTS. Furthermore, it may contribute to reduce outpatient visits, health costs and work absenteeism.

To investigate the performance and safety of the medical device eCoin™ for the treatment of refractory LUTS in patients with MS over a period of 6 months.

DETAILED DESCRIPTION:
This is a prospective, interventional, single arm, self-controlled pilot study in patients with multiple sclerosis and OAB symptoms with a 6-month treatment period of posterior tibial nerve stimulation with the medical device eCoin.

It is a pilot study to explore the effectiveness and safety of using this device to treat MS patients with OAB in daily clinical practice in. Based on feasibility considerations, we plan to include approximately 20 patients.

It consists of:

1. wash-out period from PTNS treatment of at least 2 months;
2. baseline assessments;
3. implantation of eCoin;
4. system activation; and
5. treatment and follow-up visits for a 6-month period post implant activation. Seven Visits are foreseen during the trial.

ELIGIBILITY:
Main Inclusion Criteria:

* Diagnosis of MS according to MacDonald (2011);
* Clinical stability over the past 6 months (no relapses or EDSS progression over the last 6 months);
* One or more of: urinary frequency greater than 8 times/24 hours, urinary urge incontinence at least 2 episodes in 24 hours on 3-day voiding diary
* Urodynamic diagnosis of detrusor over-activity (DOA) and / or detrusor-sphincter dyssynergia (DSD);
* Previous failure of conservative treatments (challenge over ≥6 months) i.e. lifestyle modification-fluid consumption, behavioural modification, and pharmacological therapy and stable OAB medications for at least 30 days or intolerance to pharmacological therapy (side effect);
* Positive response to ongoing PTNS treatment defined as ≥50% reduction in urinary frequency, and/or ≥50% fewer incontinence episodes, or a return to normal voiding frequency [<8 voids/day], based on retrospective diary review;
* Competent sphincter mechanism and normally functioning upper urinary tract;
* Leg circumference in the range of 20-30 cm at implantation site;
* Ability to comply with study requirements;
* Having provided written informed consent

Main Exclusion Criteria:

* Participation in another study with any investigational drug or device within the past 90 days;
* Any metal implant in the area of eCoin implantation site;
* Anatomical defects that preclude use of the device;
* Treatment with botulinum toxin injections, urinary incontinence surgery or implantation of artificial graft material, spinal or genitourinary surgery, abdominoperineal resection of the rectum or radical hysterectomy (female)/ prostatectomy (male) within the last 6 months;
* Previous treatment with sacral neuromodulation;
* Diagnosis of pelvic pain disorders, stress incontinence, current urinary tract infection, urinary stone and/or urinary tract malignancy; cystocele, enterocele or rectocele of grade 3 or 4;
* Previous or current pelvic radiotherapy and/or chemotherapy;
* Severe uncontrolled diabetes;
* Pregnant or lactating women or women planning a pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in bladder volume (mL) | Baseline and Week 24
  The patients will have their bladder filling volume measured during a urodynamic exam.
Change from baseline of detrusor pressure amplitude (cmH2O) | Baseline and Week 24
  The patients will have their detrusor pressure measured during an urodynamic exam.

SECONDARY OUTCOMES:
Change from baseline of cystometric capacity (mL) | Baseline and Week 24
  The patients will have their cystometric capacity measured during an urodynamic exam.
Change from baseline of bladder compliance (mL/cmH2O) | Baseline and Week 24
  The patients will have their bladder compliance assessed during an urodynamic exam.
Change from baseline of maximum detrusor pressure (cmH20) during storage phase | Baseline and Week 24
  The patients will have their maximum detrusor pressure during storage phase measured during an urodynamic exam.
Change from baseline of maximum detrusor pressure (cmH20) during voiding phase | Baseline and Week 24
  The patients will have their maximum detrusor pressure during voiding phase measured during an urodynamic exam.
Change from baseline of voided urine volume (mL) | Baseline and Week 24
  The patients will have their voided urine volume measured during an urodynamic exam.
Change from baseline of maximum urine flow rate (mL/s) | Baseline and Week 24
  The patients will have the maximum urine flow rate measured during an urodynamic exam.
Change from baseline of post void residual urine (mL) | Baseline and Week 24
  The patients will have the post void residual urine measured during an urodynamic exam.
Change from baseline of pelvic floor electromyographic activity | Baseline and Week 24
  The patients will have presence or absence of pelvic floor activity recorded during an urodynamic exam.
Change from baseline of vesico-uretero-renal reflux | Baseline and Week 24
  The patients will have presence or absence of vesico-uretero-renal reflux assessed during an urodynamic exam.
Change from baseline to 4, 12, and 24 weeks of bladder voiding assessed by means of a 3-day voiding diary | Baseline and Week 4, 12, 24
  The patients will self-record their bladder voiding during three consecutive days at each time point including the number of voids/day, volume voided/void, number of leaks per day, degree of urgency prior to void (none, mild, moderate, severe, incontinence), number of self-catheterization needed through the day.
Change from baseline to 4, 12, and 24 weeks of overactive bladder symptoms scores using the short form of the overactive bladder questionnaire OAB-q | Baseline, Week 4, 12, 24
  The patients will rate their overactive bladder symptoms using the OAB-qSF questionnaire. It is self-administered and asks about how much a patients is bothered by selected bladder symptoms. It contains 6 questions about symptom severity and 13 on coping, sleeping, social life each to be rated on a 6-point scale (none of the time, a little of the time, some of the time, a good bit of the time, most of the time, all of the time). Symptom severity ranges from 6 (not bothered) to 36 (extremely bothered), impact on health related quality of life ranges from 13 (not bothered) to 78 (extremely bothered).
Change from baseline to 4, 12, and 24 weeks of MSQOL54 scores. | Week -8, 4, 12, 24
  The patients will assess their health related quality of life using the short form of the MSQOL 54 questionnaire. This is a self-administered multidimensional questionnaire on health-related quality of life with generic and multiple sclerosis specific questions on physical and mental health. The summary scores are derived from 12 subscales (physical function, physical role limitations, emotional role limitations, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, sexual function). A low score indicates bad quality of life, a higher score improved quality of life (range 0-100).
Treatment satisfaction, as measured on a composite visual analogue scale (VAS) score ranging from 0-100 | Week 24
  The patients will mark a point on a 100 mm long line with a pencil to indicate their treatment satisfaction. 0 (not satisfied at all), 100 (very satisfied).
Incidence of adverse events | Week 0, 5, 12, 24
  Number and proportion of patients experiencing device related adverse events during the study period will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Chiara Zecca, PD, MD, Study Director — Ospedale Regionale di Lugano
Locations (1):
- Ospedale Regionale di Lugano, Neurocenter of Southern Switzerland, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No